CLINICAL TRIAL: NCT01019668
Title: Central Serous Chorioretinopathy Treated by Modified Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Cheng-Kuo Cheng, Assistant professor and attending physician of Ophthalmology, Shin-Kong Wu Ho-Su Memorial Hospital, School of Medicine, Fu-Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKH-8302-98-DR-27
Record Dates: First submitted 2009-11-19; First posted 2009-11-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Central Serous Chorioretinopathy
Keywords: chorioretinopathy; photodynamic therapy; reduced fluence; reduced dose
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- verteporfin PDT, half-dose (Active Comparator): use different modification of verteporfin PDT to treat prolonged unresolved central serous chorioretinopathy
  Interventions: Drug: Verteporfin PDT, half-dose; Drug: verteporfin PDT, half-fluence
- verteporfin PDT, half-fluence (Active Comparator): use different modification of verteporfin PDT to treat prolonged unresolved central serous chorioretinopathy
  Interventions: Drug: Verteporfin PDT, half-dose; Drug: verteporfin PDT, half-fluence

INTERVENTIONS:
Drug: Verteporfin PDT, half-dose — half the regular dose or half the regular laser fluence to treat prolonged unresolved CSCR
  Other Names: visudyne
Drug: verteporfin PDT, half-fluence — half the regular dose or half the regular laser fluence to treat prolonged unresolved CSCR
  Other Names: visudyne

SUMMARY:
The purpose of this study is to evaluate the effectiveness as well as the detrimental influence of half-dose and half-fluence modification of verteporfin photodynamic therapy (PDT) for the treatment of prolonged unresolved central serous chorioretinopathy (CSCR).

DETAILED DESCRIPTION:
Purpose:

to evaluate the effectiveness as well as the detrimental influence of half-dose and half-fluence modification of verteporfin PDT for the treatment of prolonged unresolved Central Serous Chorioretinopathy (CSCR).

Study Design and Patient Recruitment:

This study was a prospective, randomized, consecutive, open-labeled, comparative interventional case series. Patients with symptomatic acute or chronic CSC of 3 weeks or more duration were recruited. Patients were offered treatment if they had worsening of symptoms or no subjective improvement since the onset of the CSC. Inclusion criteria included 1) patients with best-corrected visual acuity (BCVA) of 20/400 or better; 2) presence of subretinal fluid (SRF) and/or serous pigment epithelial detachment (PED) involving the fovea on optical coherence tomography (OCT); 3) presence of active angiographic leakage in fluorescein angiography (FA) caused by CSC but not CNV or other diseases; and 4) abnormal dilated choroidal vasculature and other features in ICGA consistent with the diagnosis of CSC. Patients who received previous PDT or focal thermal laser photocoagulation for the treatment of CSC or had evidence of CNV, polypoidal choroidal vasculopathy, or other maculopathy on clinical examination, FA, or ICGA were excluded. Informed consent was obtained from all subjects. 12 patients in each group were planned to recruit in each group.

Modified Photodynamic Therapy with Half Dosage:

The Half Dosage PDT protocol for CSC was performed using half the normal dose of verteporfin (Visudyne, Novartis AG, Bülach, Switzerland) i.e., 3 mg/m2 infusion of verteporfin with a rationale that using lower dosage has less collateral damaging effects to the retina and choroid. Verteporfin was infused over 10 minutes followed by delivery of laser at 692 nm at 15 minutes from the commencement of infusion to target the area of choroidal dilation and hyperpermeability. Earlier laser application allowed less drug accumulation at the RPE layer and less drug less toxicity at the RPE. A total light energy of 50 J/cm2 over 83 seconds was delivered to the area of choroidal hyperperfusion as observed in ICGA instead of the angiographic leakage sites shown in FA. Only the area of choroidal vascular abnormality that was supposed to cause the serous detachment involving the macula was considered to be treated. To avoid overtreatment on the choroidal vasculature in causing choroidal ischemia, the laser spot size was set at a maximum of 4,500 µm. This restriction in laser spot size is adequate, from our previous report, to reverse the serous macular detachment by reducing the choroidal extravascular leakage and sub-RPE hydrostatic pressure at the macular area. In patients with bilateral CSC, only one eye was recruited for the study, and the eye with thicker central retinal thickness on OCT was chosen. After treatment, patients were given protective spectacles and instructed to avoid strong light for 3 days.

Modified Photodynamic Therapy with Half fluence:

The Half fluence PDT protocol for CSC was performed using half the normal duration of verteporfin laser time (Visudyne, Novartis AG, Bülach, Switzerland) All patients received a bolus infusion of 6 mg/m2 body surface area over 1 minute. Patients were assigned to treatment protocols, using a fluence of 25 J/cm2. In the 25-J/cm2 group, patients received an irradiance of 600 mW. Depending on the irradiance, the time of photosensitization was 42 seconds. A total light energy of 25 J/cm2 over 42 seconds was delivered to the area of choroidal hyperperfusion as observed in ICGA instead of the angiographic leakage sites shown in FA. Only the area of choroidal vascular abnormality that was supposed to cause the serous detachment involving the macula was considered to be treated. To avoid overtreatment on the choroidal vasculature in causing choroidal ischemia, the laser spot size was set at a maximum of 4,500 µm. This restriction in laser spot size is adequate, from our previous report, to reverse the serous macular detachment by reducing the choroidal extravascular leakage and sub-RPE hydrostatic pressure at the macular area. In patients with bilateral CSC, only one eye was recruited for the study, and the eye with thicker central retinal thickness on OCT was chosen. After treatment, patients were given protective spectacles and instructed to avoid strong light for 3 days.

Documentation:

Patients were seen for regular follow-up visits within 1 week before and at day 1, week 1, week 4, and month 3 after treatment. A standardized evaluation was performed at each visit including best corrected visual acuity according to the guidelines of the Early Treatment Diabetic Retinopathy Study (ETDRS), confocal scanning laser fluorescein angiography (FA), ICGA (Heidelberg Engineering, Dossenheim, Germany), fundus photography, and a complete eye examination. Selected patients were imaged with optical coherence tomography (OCT).

The main outcome measures were choroidal perfusion changes, as documented by early and late ICGA. A PDT-induced increase in collateral leakage area seen by late FA 1 day after PDT was defined as a secondary outcome, as was primary CNV closure documented by early FA. Best-corrected visual acuity was documented for safety evaluation. Data were statistically analyzed with the Wilcoxon signed-rank and Wilcoxon rank sum tests. Statistical significance was defined as P <0.05.

Procedures for Evaluation:

The Image J, (software ; NIH, USA), an imaging software developed for analysis and visualization of images obtained with grayscale photograph, was used forplanimetric evaluation of the area of hypofluorescence detected by ICGA and the area of PDT-induced leakage seen on FA. Choriocapillary hypoperfusion and nonperfusion were graded according to a scale. Angiographies were evaluated by two masked readers, and planimetricand grading results of both readers were averaged.

Follow-Up Examinations:

Patients were assessed at baseline and followed at day 1, 7, 30, 90 and 180 after PDT. At the baseline and post-PDT visits, BCVA was measured by certified optometrists with the Early Treatment Diabetic Retinopathy Study (ETDRS) logarithm of the minimum angle of resolution (logMAR) chart at 4 m or Snellen chart at 6 m being converted to logMAR equivalent for analysis. OCT recordings were performed using an OCT 3 machine (StratusOCT, Carl Zeiss Meditec Inc., Dublin, CA). Both vertical and horizontal scans of 6.0 mm centered on the fovea were obtained for measurement of central foveal thickness. OCT central foveal thickness was measured manually using the retinal thickness mode and is defined as the distance between the inner surface of the RPE and the inner surface of the neurosensory retina at the fovea. FA and ICGA were performed in all patients at baseline, month 1, and 3 after PDT. Additional FA and ICGA were carried out in patients with persistence or recurrence of CSC during the follow-up period. CSC was classified according to FA findings into two groups: 1) chronic CSC with serous retinal detachment and focal leakage (Group 1); or 2) chronic CSC with diffuse leakage that had an RPE transmission defect in early phase and diffuse angiographic leakage in mid to late phases (Group 2). Features of CSC in ICGA were delineated according to the original descriptions.

Data Analysis:

The main outcome measures of the study included the serial changes in logMAR BCVA and OCT central foveal thickness. Other outcome measures included complications and FA and ICGA changes during the follow-up period. Serial comparisons of mean logMAR BCVA and OCT central foveal thickness were performed using the nonparametric Wilcoxon-signed rank test and two-tailed t-test, respectively. Categorical variables were analyzed using the chi-square test and Fisher exact test. Statistical analysis was performed using SPSS and a P value of <=0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with best-corrected visual acuity (BCVA) of 20/200 or better
* Presence of subretinal fluid (SRF) and/or serous pigment epithelial detachment (PED) involving the fovea on optical coherence tomography (OCT)
* Presence of active angiographic leakage in fluorescein angiography (FA) caused by CSC but not CNV or other diseases
* Abnormal dilated choroidal vasculature and other features in ICGA consistent with the diagnosis of CSC.

Exclusion Criteria:

* Patients who received previous PDT or focal thermal laser photocoagulation for the treatment of CSC.
* Patients had evidence of CNV, polypoidal choroidal vasculopathy, or other maculopathy on clinical examination, FA, or ICGA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of both modification for the treatment of chronic CSCR Fluorescent leakage as regards to BCVA OCT changes | within 6 months

SECONDARY OUTCOMES:
Detrimental influence on choroidal perfusion Represented by the decrease of fluorescent intensity In ICGA | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Kuo Cheng, MD, Principal Investigator — Shin-Kong Wu Ho-Su Memorial Hospital, School of Medicine, Fu-Jen Catholic University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203